CLINICAL TRIAL: NCT07031700
Title: A Multicenter, Single-Arm, Open-Label, Phase II Trial of Mosunetuzumab in Combination With Tislelizumab for Relapsed/Refractory Follicular Lymphoma (r/r FL)
Brief Title: A Multicenter, Single-Arm, Open-Label, Phase II Trial of Mosunetuzumab in Combination With Tislelizumab for r/r FL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Director of lymphoma department, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-RR-MOS01
Record Dates: First submitted 2025-03-11; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy of Mosunetuzumab and Tislelizumab (Experimental)
  Interventions: Drug: Mosunetuzumab; Drug: Tislelizumab

INTERVENTIONS:
Drug: Mosunetuzumab — * Cycle 1: Day 1: 1 mg; Day 8: 2 mg; Day 15: 30 mg
  * Cycles 2-8: 30 mg every 3 weeks
  * Cycles 9-17: 30 mg every 3 weeks (if applicable） A treatment cycle is 21 days. Patients achieving complete remission (CR) by cycle 8 will stop treatment, while those with partial response (PR) or stable disease (SD) may continue up to 17 cycles or until disease progression or intolerable toxicity occurs.
Drug: Tislelizumab — - Cycles 2-8: 200 mg IV every 3 weeks

SUMMARY:
This is a multicenter, single-arm, open-label, investigator-initiated, phase II clinical trial designed to evaluate the feasibility, efficacy, and safety of Mosunetuzumab in combination with Tislelizumab in patients with relapsed/refractory follicular lymphoma (r/r FL).

DETAILED DESCRIPTION:
The study aims to enroll approximately 22 adult patients who have received at least two prior systemic therapies, including anti-CD20 monoclonal antibody treatment. The primary endpoint is the complete response rate (CR), while secondary endpoints include objective response rate (ORR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), and safety assessment. The trial will be conducted at multiple centers in China, with an estimated study duration from May 2025 to May 2027.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age ≥18 years.
3. Histologically confirmed relapsed/refractory follicular lymphoma (r/r FL).
4. Received at least two prior systemic therapies, including anti-CD20 monoclonal antibody therapy.
5. ECOG performance status 0-1.
6. Expected survival ≥12 weeks.
7. Measurable disease (longest diameter >1.5 cm).
8. Adequate organ function:

   * Hepatic function: Total bilirubin ≤1.5×ULN; AST/ALT ≤3×ULN.
   * Hematologic function: ANC ≥1.5 × 10⁹/L; Platelets ≥75,000/μL; Hemoglobin ≥10.0 g/dL.
   * Renal function: Serum creatinine ≤1.5×ULN or CrCl ≥50 mL/min (Cockcroft-Gault formula).
9. Women of childbearing potential must have a negative serum pregnancy test and agree to use contraception.

Exclusion Criteria:

1. Inability to comply with study hospitalization and restrictions.
2. Active infections (including tuberculosis) or immunocompromised status.
3. Prior history of severe hypersensitivity to similar agents.
4. CNS involvement of lymphoma.
5. Pregnant or breastfeeding women.
6. Uncontrolled comorbid conditions, including cardiovascular or autoimmune diseases.
7. Receipt of live attenuated vaccines within 4 weeks before enrollment.
8. Use of systemic immunosuppressants within 2 weeks prior to first dose.
9. History of drug or alcohol abuse in the past 12 months.
10. Any condition deemed inappropriate for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
best of complete response rate (CR) | up to the end of 8/17 cycles of treatment(each cycle 21 days)
  To assess the best of complete response rate (CR) at the end of treatment of Mosunetuzumab with Tislelizumab

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of 8/17 cycles of treatment(each cycle 21 days)
  Objective Response Rate is defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) after treatment with Mosunetuzumab and Tislelizumab, as assessed according to Lugano 2014 criteria.
Duration of Response (DoR) | up to 2 years
  Duration of Response is defined as the time from the first documentation of objective response (CR or PR) to the first documentation of disease progression or death from any cause, whichever occurs first. Response will be assessed per Lugano 2014 criteria.
Progression-free survival (PFS) | Assessed every 3 months during follow-up, up to 2 years
  Progression-Free Survival is defined as the time from initiation of study treatment to disease progression or death from any cause, whichever occurs first.
OS | Assessed every 3 months during follow-up, up to 2 years
  Overall Survival is defined as the time from initiation of study treatment to death from any cause.

OTHER OUTCOMES:
Identification of candidate biomarkers associated with treatment response based on RNA-seq and/or whole exome sequencing (WES) data | up to 2 years
  Tumor and/or blood samples will be collected at baseline and during treatment. RNA sequencing (RNA-seq) and/or whole exome sequencing (WES) will be performed to identify gene expression signatures, somatic mutations, or pathway alterations that correlate with clinical response (e.g., CR/PR vs. SD/PD) to the combination therapy of Mosunetuzumab and Tislelizumab.

IPD SHARING:
Plan to Share IPD: No